CLINICAL TRIAL: NCT03260413
Title: Quantifying the Burden of Hospitalizations for Pneumonia Among Children in Rural
Brief Title: Pneumonia Chart Review Cambodia
Status: Withdrawn | Type: Observational
Why Stopped: Could not get IRB approval
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000091
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pneumonia cases: Children between the ages of 1 month through 5 years of age who are admitted to Chenla Children's Healthcare between opening of the hospital (mid-2017) and early February 2018 for pneumonia and respiratory distress.

SUMMARY:
This study aims to answer the question of what is the burden of lower respiratory disease (pneumonia) among children ages 1 month to 5 years of age in rural Cambodia. The primary objective will be to quantify the prevalence of severe pneumonia at Chenla Children's Healthcare, a hospital in the rural town of Kratie, Cambodia. This will involve a chart review of the medical records available at Chenla Children's Healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 1 month and 5 years admitted to Chenla Children's Healthcare with at least one admitting diagnosis being pneumonia or bronchiolitis will be included.

Exclusion Criteria:

* Children who do not fall into the aforementioned age range and who do not have "pneumonia" or "bronchiolitis" as one of the admitted diagnoses.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be children between the ages of 1 month and 5 years who were admitted to Chenla Children's Healthcare with at least one admitting diagnosis being "pneumonia" or "bronchiolitis". These children will be residents of Kratie province, Cambodia. They are admitted to Chenla Children's Healthcare by way of their emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-12 (Estimated); Primary Completion 2018-03-09 (Estimated); Study Completion 2018-03-09 (Estimated)

PRIMARY OUTCOMES:
Pneumonia count | 5-6 months
  Number of admissions for pneumonia to Chenla Children's healthcare

IPD SHARING:
Plan to Share IPD: Yes
The data from this chart review will be used to inform baseline information of a larger study that is currently in the planning stages. All investigators participating in this chart review are also investigators in this larger study. Information from this chart review will only be accessed by investigators participating in this larger study and by no one outside of this larger study.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: The data will become available by March 10, 2018. It will be available for 4 years.